CLINICAL TRIAL: NCT04622956
Title: GVHD Prophylaxis With Methotrexate and Cyclosporine in Haploidentical Stem Cell Transplantation Using Posttransplant Cyclophosphamide in Hematologic Malignancies: Phase I/II Trial
Brief Title: GVHD Prophylaxis With Methotrexate in Haploidentical HCT Using Posttransplant Cyclophosphamide
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 30802020.7.1001.0068
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Graft Vs Host Disease; Hematopoietic Neoplasm
Keywords: Methotrexate; Post-transplant cyclophosphamide; Cyclosporine; Haploidentical; Hematopoietic cell transplantation
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase I / II multicenter open-label clinical trial with prospective nonrandomized arm and historical control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): GVHD prophylaxis will consist of high-dose PTCy (50 mg/kg i.v. on days +3 and +4) with mesna, cyclosporine (initiated on day +5) and methotrexate i.v (see doses on the right). Cyclosporine will be dosed with a target trough of 200 to 250 ng/mL and discontinued without taper at D+60 (if bone marrow graft) or until D+90 (is peripheral blood graft), unless acute GVHD is present. Filgrastim will be administered from day +5 until neutrophil recovery to ≥ 1,000/mcL for 3 days.
  Interventions: Drug: Methotrexate Injectable Solution
- Control Group (No Intervention): GVHD prophylaxis will consist of high-dose PTCy (50 mg/kg i.v. on days +3 and +4) with mesna, cyclosporine (initiated on day +5) and mycophenolate mofetil (15 mg/kg/dose p.o. t.i.d. initiated on day +5). Cyclosporine will be dosed with a target trough of 200 to 250 ng/mL and discontinued without taper at D+60 (if bone marrow graft) or until D+90 (is peripheral blood graft), unless acute GVHD is present.

INTERVENTIONS:
Drug: Methotrexate Injectable Solution — Phase 1:
  * Level -1: Methotrexate 7.5 mg/m2 on D+6 and D+9*. Level -1 will be explored only if the starting dose is too toxic (reduced dose).
  * Level 0 [Starting Dose]: Methotrexate 10 mg/m2 on D+6 and 7.5 mg/m2 on D+9
  * Level +1: Methotrexate 10 mg/m2 on D+6 and D+9
  * Level +2: Methotrexate 15 mg/m2 on D+6 and 10 mg/m2 on D+9
  Phase 2: dose determined in the phase 1 trial
  Other Names: Fauldmetro [Libbs]
  Arms: Experimental

SUMMARY:
Allogeneic hematopoietic cell transplantation (HCT) is an important therapeutic strategy for many malignant and benign hematologic diseases. Haploidentical HCT has been increasingly used in patients lacking a HLA-matched donor due to its prompt availability, possibly lower cost and results comparable with other donor types. Graft-versus-host disease (GVHD) is the main cause of morbidity and mortality after HSCT, and prophylactic strategies are routinely used. In the context of haploidentical HCT, posttransplant cyclophosphamide plus cyclosporine and mycophenolate mofetil (MMF) is the most common platform used in Brazil. Data comparing MMF and methotrexate (MTX) as GVHD prophylaxes have proved controversial in other donor types, yet some large studies have showed that MTX is associated with lower risk of GVHD and improved long-term outcomes. Moreover, it is known that MMF is a potent inhibitor of natural killer (NK) cells, possibly interfering with the graft-versus-leukemia effect in haploidentical HCT. Given the possible advantages and the absence of consistent evidence regarding safety, efficacy and ideal dosage of MTX as GVHD prophylaxis in this setting, we propose a phase I / II study evaluating this drug in adult patients with hematologic malignancies undergoing haploidentical HCT with posttransplant cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia and chronic myeloid leukemia in complete morphologic remission, myelodysplastic syndrome with less than 10% in bone marrow or peripheral blood, Ph-negative acute lymphoblastic leukemia in complete morphologic remission, chemosensitive Hodgkin lymphoma or non-Hodgkin lymphoma in at least partial remission
* Donor type: haploidentical related donor
* Graft source: bone marrow or peripheral blood
* Recipients of non-myeloblative or myeloablative intensity conditioning
* Left Ventricle Ejection fraction > 40%
* Estimated creatinine clearance > 40 mL/min
* Adjusted DLCO ≥ 40% and FEV1 ≥ 40%
* Total bilirubin < 2x ULN e ALT/AST < 2.5x ULN

Exclusion Criteria:

* Prior allogeneic transplant
* Ex-vivo graft manipulation (T-cell-depleted or CD34-selected grafts)
* Use of alemtuzumab or anti-thymocyte globulin
* KPS < 70%
* Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment
* Pregnant or lactating women
* Patients seropositive for human immunodeficiency virus (HIV) or active hepatitis B or C infection by PCR
* Presence of fluid collection (ascites, pleural or pericardial effusion) that may interfere with methotrexate clearance or make methotrexate use contraindicated
* Patients with a serious medical or psychiatric illness likely to interfere with participation in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Methotrexate dose to be used in the phase 2 (Phase 1) | Day 30
  The methotrexate dose to be used in the subsequent phase 2 will be equal to or lower than the maximum tolerated dose (MTD). MTD will be considered exceeded if at least 2 out of 6 subjects on a certain dosing level develop dose-limiting toxicity (DLT). DLT consists of gastrointestinal tract perforation, mediastinitis, airway obstruction requiring orotracheal intubation, severe gastrointestinal bleeding (without evidence of GVHD), graft failure, or hyperbilirubinemia or increase in alanine transaminase [ALT] / aspartate transaminase [AST] levels > 5x the upper limit of normal.
GVHD-free, relapse-free survival (Phase 2) | Day 365
  Relapse, grade 3-4 GVHD and 2014 NIH Chronic GVHD will be considered events, and non-relapse related mortality will be a competing event.

SECONDARY OUTCOMES:
Overall survival | Day 365
  Time to death
Cumulative incidence of neutrophil and platelet engraftment | Day 30
  Neutrophil engraftment will be the first of three consecutive daily absolute neutrophil counts > 500 / mcL after transplantation. Disease relapse will be a competitive event. Platelet engraftment will be considered as the first of seven daily consecutive platelet counts > 20,000 / mcL without transfusion support. Disease relapse will be a competitive event.
Cumulative incidence of graft failure | Day 30
  Time to primary or secondary graft failure. Primary graft failure will be defined as failure to reach neutrophils > 500 / mcL for three consecutive days or donor chimerism <5% in any hematopoietic compartment (lymphocyte chimerism or total bone marrow / peripheral blood chimerism) and requiring additional hematopoietic cells. Secondary graft failure will be defined as the need for additional hematopoietic cells due to declining hematopoietic recovery in a patient with previous neutrophil engraftment.
Cumulative incidence of grade II-IV acute GVHD | Day 100
  Time to onset of grade II-IV acute GVHD according to the MAGIC criteria. Death without previous acute GVHD will be a competing event.
Cumulative incidence of grade III-IV acute GVHD | Day 100
  Time to onset of grade III-IV acute GVHD according to the MAGIC criteria. Death without previous acute GVHD will be a competing event.
Cumulative incidence of non-relapse/progression related mortality | Day 365
  Time to onset of disease relapse or progression (imaging, morphologic or molecular). Non-relapse related mortality will be a competing event.
Cumulative incidence of Chronic GVHD | Day 365
  Time to onset of 2014 NIH Chronic GVHD. Non-relapse related mortality will be a competing event.
Change in 36-Item Short Form Health Survey (SF-36) | Baseline, Days 30, 90, 180, and 365
  Change in mean subscale response of the SF-36 Survey version 2.0 (Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Energy/fatigue, Emotional well-being, Social
Change in the Functional Assessment of Cancer Therapy (FACT)-Bone Marrow Transplantation (BMT) Survey | Baseline, Days 30, 90, 180, and 365
  Change in mean subscale response of the FACT-BMT survey
Frequency of Grade 3-5 adverse events | Day 30
  Adverse events will be classified according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), Version 5.0
Change in Natural Killer cell function [% activity] | Days 30, 90, and 180
Change in lymphocyte subsets [absolute number/mcL] | Days 30, 90, and 180
Cumulative incidence of CMV and EBV reactivation | Day 100
Change in bone marrow or peripheral blood donor chimerism [%] | Days 30, 90, and 180
Change in mean free mycophenolic acid and mycophenolic acid glucuronide level [mcg/mL] on peripheral blood (controls only) | Days 12 and 19

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Fatobene, MD, Principal Investigator — Hospital das Clínicas da Universidade de São Paulo
Locations (4):
- Brazil (4):
  - Instituto Nacional de Câncer José Alencar Gomes Da Silva - Inca, Rio de Janeiro, Rio de Janeiro
  - Centro de Hematologia e Hemoterapia - HEMOCENTRO, Campinas, São Paulo
  - Hospital Amaral Carvalho / Fundação Dr. Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clinicas da Universidade de Sao Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No